CLINICAL TRIAL: NCT05018767
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Aging Frailty
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Intravenous Infusion for Aging Frailty
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-11-ATG-12-01
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Frailty
Keywords: Frailty; stem cell treatment; Anti Aging
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of Aging Frailty

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Aging Frailty. This patient funded trial aims to study the safety and efficacy of intravenous infusion of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of Frailty. Patients with Frailty will receive a single intravenous infusion of UC-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Aging Frailty
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (3):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Athens Beverly Hills Medical Group, Glyfada, Athens, Greece
- Artros, Ljubljana, Slovenia, Slovenia

REFERENCES:
- [Background] Tompkins BA, DiFede DL, Khan A, Landin AM, Schulman IH, Pujol MV, Heldman AW, Miki R, Goldschmidt-Clermont PJ, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Da Fonseca M, Golpanian S, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Green G, Oliva AA, Hare JM. Allogeneic Mesenchymal Stem Cells Ameliorate Aging Frailty: A Phase II Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1513-1522. doi: 10.1093/gerona/glx137. PMID 28977399
- [Background] Golpanian S, DiFede DL, Khan A, Schulman IH, Landin AM, Tompkins BA, Heldman AW, Miki R, Goldstein BJ, Mushtaq M, Levis-Dusseau S, Byrnes JJ, Lowery M, Natsumeda M, Delgado C, Saltzman R, Vidro-Casiano M, Pujol MV, Da Fonseca M, Oliva AA Jr, Green G, Premer C, Medina A, Valasaki K, Florea V, Anderson E, El-Khorazaty J, Mendizabal A, Goldschmidt-Clermont PJ, Hare JM. Allogeneic Human Mesenchymal Stem Cell Infusions for Aging Frailty. J Gerontol A Biol Sci Med Sci. 2017 Oct 12;72(11):1505-1512. doi: 10.1093/gerona/glx056. PMID 28444181